CLINICAL TRIAL: NCT03494036
Title: Effect of Synbiotic Supplementation on Interleukin 17 (IL-17) Level, Regulatory T-cells, Gut Permeability and Microbiota in Patient With Connective Tissue Disease
Brief Title: Effect of Synbiotic on Immune Response, Gut Permeability and Microbiota in Patient With Connective Tissue Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, alvinawidhani, Principal Investigator, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 804/UN2.F1/ETIK/2017
Record Dates: First submitted 2018-03-31; First posted 2018-04-11 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Connective Tissue Diseases
Keywords: synbiotic; probiotic; lupus; connective tissue disease
MeSH Terms: conditions — Connective Tissue Diseases | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic (Experimental): Synbiotic capsule containing 3x1.000.000.000 Colony Forming Units probiotics (Lactobacillus helveticus R0052 60%, Bifidobacterium infantis R0033 20%, dan Bifidobacterium bifidum R0071 20%) and fructooligosaccharide 80 mg. The dosage is once daily and it is given for 60 days
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Placebo Comparator): Placebo capsule containing saccharum lactis. The dosage is once daily and it is given for 60 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — capsule
  Arms: Synbiotic
Dietary Supplement: Placebo — capsule
  Arms: Placebo

SUMMARY:
This is a double blind randomized placebo controlled trial to determine the effect of synbiotic to FOXP3 regulatory T cells, IL-17, gut permeability and gut microbiota in patients with connective tissue disease. Synbiotic can increase FOXP3 regulatory T cells, decrease IL-17 and improve gut permeability and gut microbiota in patients with connective tissue disease.

DETAILED DESCRIPTION:
Study showed gut microbiota has a role in the pathogenesis of autoimmune diseases. Gut microbiota which can increase gut permeability affect the antigen presentation to the immune system. Synbiotic supplementation is expected to improve immune system, gut permeability, and gut microbiota in patients with connective tissue disease.

The subjects who fulfill inclusion criteria, willing to participate and sign informed consent will be randomized into two groups: the group receiving synbiotic containing probiotic (Lactobacillus helveticus R0052 60%, Bifidobacterium infantis R0033 20%, dan Bifidobacterium bifidum R0071 20%) and 80 mg fructooligosaccharide (group I, n=23) and the group receiving placebo (group II, n=23). Both groups receive intervention for two months. Patients continue to receive their immunosuppressive drugs (corticosteroids, hydroxychloroquine, mycophenolate mofetil, azathioprine, or cyclosporine).

Percentage of FOXP3 Regulatory T-cells, serum IL-17, zonulin, high sensitivity C-reactive protein, and gut microbiota are evaluated at the beginning and at the end of the study. FOXP3 regulatory T-cell is evaluated by flowcytometry. Serum IL-17 and zonulin are measured by ELISA. Gut microbiota is evaluated using 16s ribosomal RNA gene next generation sequencing. The DNA from the stool is isolated by DNA stool mini kit (QIAamp).

The results are presented in mean ± standard deviation, median (IQR 25-75%) and n (%). The Kolmogorov-Smirnov test is used to determine the normality of the data, assuming the normality of the data is fulfilled if p> 0.05. Bivariate analysis uses paired T test if the data has normal distribution. If the distribution is not normal, Wilcoxon test will be used. Differences are said to be significant when the value of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with connective tissue disease
* has gastrointestinal symptoms (abdominal pain, diarrhea, constipation, or bloating)
* age between 18-60 years old

Exclusion Criteria:

* pregnant or breastfeeding
* acute infection
* on antibiotic treatment
* taking yoghurt or probiotic supplementation in the last 3 weeks before recruitment
* taking corticosteroid more than 20 mg prednison a day or equal\
* refuse to join the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
FOXP3 regulatory T cell | 2 months
  change in the percentage of FOXP3 regulatory T cell

SECONDARY OUTCOMES:
IL-17 | 2 months
  change in the serum IL-17 level
zonulin | 2 months
  change in the serum zonulin level
gut microbiota | 2 months
  change of the profile of gut microbiota

CONTACTS AND LOCATIONS:
Overall Officials: alvina widhani, MD, Principal Investigator — Faculty of Medicine University of Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, Indonesia